CLINICAL TRIAL: NCT02144519
Title: Nutrition and Physical Activity Policies, Obesogenic Behaviors and Weight Outcomes
Brief Title: Physical Activity and Nutrition Intervention in Afterschool Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Beets, Dr. Michael W. Beets, PhD, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R01HL112787-01A1 (NIH); 1R01HL112787-01A1 (NIH)
Record Dates: First submitted 2014-05-13; First posted 2014-05-22 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Diet, Healthy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Intervention (Experimental): Over the 3 year project, this arm receives the Healthy Eating and Physical Activity intervention after year 1 (baseline) for a total of 2 years (year 2 and 3).
  Interventions: Behavioral: Healthy Eating and Physical Activity
- Delayed Intervention (Experimental): Over the 3 year project, this arm serves as the no treatment control/comparison group for year 1 and 2 (2 years of baseline) and receives the Healthy Eating and Physical Activity intervention in year 3 for a total of 1 year.
  Interventions: Behavioral: Healthy Eating and Physical Activity

INTERVENTIONS:
Behavioral: Healthy Eating and Physical Activity — Create partnerships with ASPs to help facilitate changes in programming to meet the National Afterschool Alliance's HEPA Standards.
  Other Names: HEPA

SUMMARY:
The investigators long-term goal is to advance the adoption and successful implementation of policies that promote PA and nutrition in after school programs (ASP) nationwide. The investigators objective here is two fold. First, the investigators will test the effectiveness of two promising strategies designed to 1) increase the amount of PA children accumulate while attending an ASP and 2) promote changes in the nutritional quality of the snacks served. This represents a fundamental step in establishing practice-based guidelines (best practices) for the uptake and achievement of public health policy goals (CA and Harvard). Second, the investigators will examine the barriers and facilitators to implementing these strategies. The expected outcome of this study is evidence supporting best practices for ASPs to employ to meet policy goals.

DETAILED DESCRIPTION:
The investigators will use a 3-year delayed treatment, cluster randomized controlled trial design with 20 ASPs that serve mostly low-income and minority children (approximately 1300 children ages 6-12yrs) in Columbia, SC and address the following specific aims: Aim 1. Evaluate the impact of a staff-level intervention, a professional development training program focused on core competencies to promote physical activity, on children's physical activity levels; Aim 2. Evaluate the impact of a site-level intervention, a snack modification program that includes a discount buying program, on the quality of snacks served and consumed; and Aim 3. Evaluate the implementation of the staff-level and site-level interventions and identify organizational, staff, and setting characteristics that influence the process of implementing these strategies.

ELIGIBILITY:
Inclusion Criteria:

Programs that:

* Operate immediately after the school day
* Operate every day of the school year for a minimum of 2 hours
* Serve a minimum of 30 children of elementary age (6-12 years)
* Operate in a school, community or faith Setting
* Provide a snack
* Provide homework assistance/completion time
* Provide enrichment
* Provide opportunities for physical activity
* All children enrolled, staff, and afterschool program (ASP) leaders in the ASPs were eligible to participate in the study.

Exclusion Criteria:

* Programs that:
* Were singularly focused
* Programs that were physical activity focused

Children that:

* Have any physical and/or orthopedic impairment that would limit a child's ability to participate in regular physical activity.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2635 (Actual)
Dates: Start 2012-08; Primary Completion 2015-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Beets, PhD, Principal Investigator — University of South Carolina

REFERENCES:
- [Derived] Beets MW, Weaver RG, Turner-McGrievy G, Huberty J, Ward DS, Pate RR, Freedman D, Hutto B, Moore JB, Bottai M, Chandler J, Brazendale K, Beighle A. Physical activity outcomes in afterschool programs: A group randomized controlled trial. Prev Med. 2016 Sep;90:207-15. doi: 10.1016/j.ypmed.2016.07.002. Epub 2016 Jul 7. PMID 27397608
- [Derived] Beets MW, Weaver RG, Turner-McGrievy G, Huberty J, Ward DS, Freedman D, Hutto B, Moore JB, Beighle A. Making Healthy Eating Policy Practice: A Group Randomized Controlled Trial on Changes in Snack Quality, Costs, and Consumption in After-School Programs. Am J Health Promot. 2016 Sep;30(7):521-31. doi: 10.4278/ajhp.141001-QUAN-486. Epub 2016 Jun 17. PMID 26158679
- [Derived] Beets MW, Weaver RG, Turner-McGrievy G, Huberty J, Ward DS, Pate RR, Freedman D, Hutto B, Moore JB, Beighle A. Making policy practice in afterschool programs: a randomized controlled trial on physical activity changes. Am J Prev Med. 2015 Jun;48(6):694-706. doi: 10.1016/j.amepre.2015.01.012. PMID 25998921

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Differences between the total number of children with outcome measures collected and the number of children measured at baseline is due to the use of a repeated-cross sectional design where a total of 2635 unique children were measured across 3 years and a subset with 2 or more years participating in outcome measurements.
Units Other Than Participants: Afterschool Programs
Period: Year 1
Arm/Group | Immediate Intervention | Delayed Intervention
Started | 895; 10 Afterschool Programs | 870; 10 Afterschool Programs
Completed | 895; 10 Afterschool Programs | 870; 10 Afterschool Programs
Not Completed | 0; 0 Afterschool Programs | 0; 0 Afterschool Programs
Period: Year 2
Arm/Group | Immediate Intervention | Delayed Intervention
Started | 763; 10 Afterschool Programs | 864; 10 Afterschool Programs
Completed | 763; 10 Afterschool Programs | 864; 10 Afterschool Programs
Not Completed | 0; 0 Afterschool Programs | 0; 0 Afterschool Programs
Period: Year 3
Arm/Group | Immediate Intervention | Delayed Intervention
Started | 894; 10 Afterschool Programs | 760; 10 Afterschool Programs
Completed | 894; 10 Afterschool Programs | 760; 10 Afterschool Programs
Not Completed | 0; 0 Afterschool Programs | 0; 0 Afterschool Programs

BASELINE CHARACTERISTICS:
Groups:
- Delayed Intervention: This arm served as a comparison group for the first year and received the Healthy Eating and Physical Activity intervention in year 3 along with arm 1.
  Healthy Eating and Physical Activity: Create partnerships with ASPs to help facilitate changes in programming to meet the National Afterschool Alliance's HEPA Standards.
- Immediate Intervention: This arm receives the Healthy Eating and Physical Activity intervention in ASPs intervention immediately for a full year before the delayed intervention begins. This arm gets the intervention and support for two years.
  Healthy Eating and Physical Activity: Create partnerships with ASPs to help facilitate changes in programming to meet the National Afterschool Alliance's HEPA Standards.
- Total: Total of all reporting groups
Arm/Group | Delayed Intervention | Immediate Intervention | Total
Number analyzed (Participants) | 870 | 895 | 1765
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.1 (1.8) | 7.9 (1.8) | 8.0 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 414 | 417 | 831
  Male | 456 | 478 | 934
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 421 | 578 | 999
  Black | 389 | 266 | 655
  Other | 60 | 51 | 111
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 870 | 895 | 1765
Percentage of Achieving 30min Moderate-to-Vigorous Physical Activity (MVPA) Standard via acceleromtr [Number; unit: % Achieving MVPA Standard] — All children attending an ASP on unannounced measurement days had an opportunity to wear the ActiGraph GT3X+. The accelerometers were distilled using 5-second epochs. When children arrived to a program, they were fitted with an accelerometer and the arrival time was recorded (monitor time on). Before a child departed from a program, research staff removed the belt and recorded the time of departure (monitor time off). Children wore the monitors for their entire attendance at the ASPs.
  % Achieving MVPA Standard
    Girls | 15 | 16.2 | 15.5
    Boys | 31.8 | 35.6 | 33.2

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Children Meeting Physical Activity Policy
Description: We will assess the number of children meeting the physical activity policy of 30 minutes or more of moderate-to-vigorous physical activity. The primary physical activity (PA) and sedentary behavior outcome was derived via accelerometry. All children attending an ASP on unannounced measurement days had an opportunity to wear the ActiGraph GT3X+. The accelerometers were distilled using 5-second epochs. When children arrived to a program, they were fitted with an accelerometer and the arrival time was recorded (monitor time on). Before a child departed from a program, research staff removed the belt and recorded the time of departure (monitor time off). Children wore the monitors for their entire attendance at the ASPs. Cutpoint thresholds associated with moderate and vigorous activity were used to distill the PA intensity levels and sedentary behavior. Children were considered to have a valid day of accelerometer data if their total wear time (time off minus time on) was ≥60 minutes.
Time Frame: Spring of Year 1, Year 2, and Year 3
Population: Analysis based on the percentage of children (boys and girls, separately) achieving the 30 min MVPA standard
Measure: Number; unit: Percent children achieving MVPA standard
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 1290 | 1345
Percent children achieving MVPA standard
  Year 1 - Boys: number analyzed (Participants) | 477 | 456
  Year 1 - Boys | 35.9 | 29.0
  Year 2 - Boys: number analyzed (Participants) | 452 | 443
  Year 2 - Boys | 44.2 | 29.3
  Year 3 - Boys: number analyzed (Participants) | 485 | 383
  Year 3 - Boys | 47.0 | 31.3
  Year 1- Girls: number analyzed (Participants) | 418 | 414
  Year 1- Girls | 19.1 | 13.1
  Year 2 - Girls: number analyzed (Participants) | 411 | 421
  Year 2 - Girls | 24.3 | 12.3
  Year 3 - Girls: number analyzed (Participants) | 409 | 377
  Year 3 - Girls | 21.6 | 19.1
Statistical Analysis 1: Comparison: Immediate Intervention vs Delayed Intervention; Test type: Superiority; p = 0.008, Mixed Models Analysis; Odds Ratio (OR) = 1.88, 95% CI 2-sided [1.18 to 3.00]

2. Secondary Outcome: Changes in Nutritional Quality of Snacks
Description: We will assess quality of snacks served at the ASPs in terms of number of fruits and vegetables served per week. These analyses were performed at the ASP level with a sample size of 20 (10 per arm)
Time Frame: Spring of Year 1, Year 2, and Year 3
Population: Direct observation of the number of days per week a fruit or vegetable was served
Measure: Mean (Standard Deviation); unit: Days/Week Fruit/Vegetables served
Units Other Than Participants: Afterschool Programs
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | NA | NA
Number analyzed (Afterschool Programs) | 10 | 10
Days/Week Fruit/Vegetables served
  Year 1 | 0.6 (1.6) | 0.7 (1.8)
  Year 2 | 4.1 (1.9) | 0.8 (1.8)
  Year 3 | 4.3 (1.7) | 1.7 (2.4)
Statistical Analysis 1: Comparison: Delayed Intervention; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 3.80, 95% CI 2-sided [1.45 to 9.95]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Delayed Intervention | Immediate Intervention
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No